CLINICAL TRIAL: NCT07099040
Title: IMPlementation stRategiEs for Scalability and Sustainability - Multidomain INterventions in a Structured Care Pathway to Detect and Delay Cognitive Decline in Community-dwelling Older Adults (IMPRESS-MIND2S): Pilot Test
Brief Title: Community-based Multi-domain Intervention to Detect and Delay Cognitive Decline in Community-dwelling Older Adults: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202503-0001; NICTran2023-0014 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2025-03-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Mild Cognitive Impairment (MCI)
Keywords: Multi-domain intervention; Pilot study; Community-based intervention; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Twice of physical activity at the AAC with home-based exercises once to twice a week, and once a week of cognitive activity at the AAC, with once to twice a week of home-based activity
  Interventions: Behavioral: Social support; Behavioral: Health coaching; Behavioral: Physical Activity; Behavioral: Cognitive activity
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Social support — Psychoeducation will be provided for enrolled participants and their caregivers by Community Resource, Engagement & Support Team (CREST). Visits from CREST teams will be provided on an ad hoc basis, based on older adult participants' needs and circumstances.
  Arms: Intervention
Behavioral: Health coaching — Health coaching aims to control risk factors of dementia by community nurses (CMNs) and wellbeing coordinators (WBCs). These include addressing chronic conditions and lifestyle aspects (diet, exercise, habits stress management, and sleep). Care recipients are encouraged to proactively manage their health journey and establish Specific, Measurable, Achievable, Relevant, and Time-bound (SMART) goals with the support of WBCs and CMNs. This multi-faceted approach has the potential to not only address older individuals' immediate health concerns but also foster long-term lifestyle changes. The frequency of visits are once or twice a month, depending on recipients' health status and cognitive functions.
  Flexible scheduling is based on individual needs and community nurses' usual practice at the Community Health Post at AACs.
  Arms: Intervention
Behavioral: Physical Activity — Physical Activity that focuses on improving resistance and balance for care recipients. Physical activity will be conducted 2 times/week at the Active Ageing Centres (AACs) with care recipients for a duration of 1-hour and 1-2 times/week at home.
  Arms: Intervention
Behavioral: Cognitive activity — Cognitive activity will be delivered to enrolled care recipients by Community Resource, Engagement & Support Team (CREST) and AAC staff. With the incorporation of using SilverPad as part of the cognitive activities, care recipients will undergo 1-hour weekly cognitive activity. Youth volunteers will also be engaged to help facilitate the sessions.
  This will be augmented with additional 1-2 times weekly home-based training sessions supervised by caregivers.
  Arms: Intervention

SUMMARY:
The incidence of cognitive impairment and its burden are increasing with a rapidly ageing population. In Singapore, the prevalence of dementia among older adults aged 60 and above is approximately 10%, which will translate to approximately 152,000 older adults living with dementia by the year 2030. Using 2013 data as estimates, the total annual cost of dementia was already estimated at S$532 million while cost per person was estimated at S$10,245 per annum, and a further increase in corresponding costs is expected through 2030 with the projection of increase in persons with dementia (PWDs). There is thus an urgent need for (i) effective, scalable, and sustainable interventions that are widely accessible to detect and delay cognitive decline and frailty in our community-dwelling older adults, and (ii) providing support for their caregivers. This study aims to test the feasibility of a community-based multi-domain intervention for detecting and delaying cognitive impairment for the older population.

ELIGIBILITY:
Inclusion Criteria

Older Adults:

* 60 years and older with cognitive concerns or (self-reported or observer reported),
* English and/or Mandarin speaking,
* no physical disabilities that preclude study participation,
* willing to complete all study-related activities,
* no known diagnosis of major cognitive impairment,
* able to provide consent.

Caregivers:

* 21 years and older,
* English and/or Mandarin speaking,
* able to provide consent
* have at least 6-month experience of taking care of older adults with mild cognitive impairment.

Service providers:

* 21 years and older,
* English and/or Mandarin speaking,
* able to provide consent.

Youth Volunteers:

* volunteers from Youth Corps Singapore (YCS)
* English and/or Mandarin speaking,
* able to provide assent

Exclusion Criteria:

Older adults

* Known diagnosis of moderate dementia and above,
* Montreal Cognitive Assessment (MoCA) score <18,
* Has difficulty in basic activities of daily living,
* disorders that affects safe engagement in the intervention (e.g. symptomatic cardiovascular disease, revascularization within 1 year, major depression or anxiety with ongoing treatment, underlying malignancy),
* Severe vision or hearing impairment or any other disorders preventing cooperation as judged by the study team,
* Major illness with life expectancy <6 months,
* Institutionalized,
* Planned major surgery within the duration of the multi-domain intervention,
* Physical disabilities that preclude study participation.

Caregivers:

* aged below 21 years old,
* not being the primary family caregiver of at least one older individual,
* not being able to read, write, and converse in English/Mandarin,
* their family members (older adults) have not participated in the pilot test for at least one month (1 session of cognitive activity/week, 2 sessions of physical activity/week).

Care providers:

* not working for the older population,
* Not being able to read, write, and converse in English/Mandarin,
* have not provided service during the period of the pilot test for at least one month (1 session of cognitive activity/week, 2 sessions of physical activity/week).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-08-12 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Care recipients' cognition measured by the Montreal Cognitive Assessment (MoCA) | From enrollment to the end of month 6
  The MoCA (Montreal Cognitive Assessment) scoring ranges from 0 to 30, with a higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Care recipients' physical function measured by short physical performance battery (SPPB) | From enrollment to the end of month 6
  The Short Physical Performance Battery (SPPB) assesses lower extremity function in older adults by evaluating standing balance, gait speed, and repeated chair stands, with scores ranging from 0 to 12, where higher scores indicate better function.
Care recipients' frailty measured by FRAIL scale | From enrollment to the end of month 6
  The FRAIL scale (Fatigue, Resistance, Ambulation, Illnesses, and Loss of weight) is a clinical screening tool used to identify frailty in older adults.
  Scoring breakdown:
  * Each component is scored as 0 or 1
  * Minimum total score: 0
  * Maximum total score: 5
  Higher scores indicate worse outcomes/greater frailty:
  The five components are scored as follows:
  * Fatigue: "Are you fatigued?" (Yes = 1, No = 0)
  * Resistance: "Can you climb one flight of stairs?" (No = 1, Yes = 0)
  * Ambulation: "Can you walk one block?" (No = 1, Yes = 0)
  * Illnesses: Having 5 or more illnesses (Yes = 1, No = 0)
  * Loss of weight: >5% weight loss in past 6 months (Yes = 1, No = 0)
Care recipients' health-related quality of life measured by EuroQol 5-Dimension 5-Level (EQ-5D-5L) | From enrollment to the end of month 6
  EuroQol 5-Dimension 5-Level (EQ-5D-5L)
  For the individual dimension scores (Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression):
  * Minimum value: 1
  * Maximum value: 5
  * Higher scores = Worse health outcomes
Care recipients' health state on a EuroQol Visual Analogue Scale (EQ VAS) | From enrollment to the end of month 6
  For the EuroQol Visual Analogue Scale (EQ VAS):
  * Minimum value: 0
  * Maximum value: 100
  * Higher scores = Better health outcomes
Caregivers' caregiving burden measured by Zarit burden interview (ZBI) | From enrollment to the end of month 6
  The Zarit Burden Interview-12 (ZBI-12) or Short Version of Zarit Burden Interview:
  * Minimum score: 0
  * Maximum score: 48
  * Higher scores indicate greater caregiver burden
  Scoring interpretation:
  * 0-10: No to mild burden
  * 11-20: Mild to moderate burden
  * 20: High burden
Care recipients' ability to perform more complex tasks necessary for independent living within the community - Measured by Lawton scale iADL | From enrollment to the end of month 6
  Each item in iADL is rated based on the person's ability to perform the task independently, with some versions scoring:
  0 = unable or needs help
  1 = independent
  Total scores range from 0 (low function, dependent) to 8 (high function, independent).
Feasibility outcome - Acceptability, collected from the Acceptability of Intervention Measure (AIM) | At the end of months 2, 4, and 6
  AIM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Perceived appropriateness, collected from the Intervention Appropriateness Measure (IAM) | At the end of months 2, 4, and 6
  IAM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Perceived feasibility, collected from the Feasibility of Intervention Measure (FIM) | At the end of months 2, 4, and 6
  FIM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Care recipients' perceptions of the intervention, collected from qualitative interview | Month 6
Feasibility outcome - Acceptability, collected from the Acceptability of Intervention Measure (AIM) | Month 6
  AIM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Perceived appropriateness, collected from the Intervention Appropriateness Measure (IAM) | Month 6
  IAM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Perceived feasibility, collected from the Feasibility of Intervention Measure (FIM) | Month 6
  FIM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Caregivers' perceptions of the intervention, collected from qualitative interview | Feasibility outcome - Caregivers' perceptions of the intervention, collected from qualitative interview
Feasibility outcome - Acceptability, collected from the Acceptability of Intervention Measure (AIM) | From enrollment to the end of month 6
  AIM has 4 items describing participants' acceptance of the intervention. Each item has 5 possible options, with scoring
  1. - Completely disagree
  2. - Disagree
  3. - Neither agree nor disagree
  4. - Agree
  5. - Completely agree
Feasibility outcome - Caregivers' perceptions of the intervention, collected from qualitative interview | Month 6